CLINICAL TRIAL: NCT01328704
Title: Observational Study to Evaluate Changes in Iron, Vit-D, and CRP During a Twelve to Twenty-Four Week Supervised Triathlon Training Program
Brief Title: Evaluate the Change in Iron, Vitamin D, and C-Reactive Protein Level (CRP) in a 12 to 24 Week Period
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: ARI-1390-Triathletes
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Anemia; Vitamin D Deficiency
Keywords: Iron deficiency; Vitamin D deficiency; Anemia; Athletes; Triathletes; Triathlon
MeSH Terms: conditions — Anemia; Vitamin D Deficiency; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained three times throughout the course of the subject's involvement in the study: baseline, 3 months, and 6 months.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Triathletes: Group of individuals who are participating in a triathlon training program at the Avera Sports Institute

SUMMARY:
The purpose of this study is to observe changes in iron status and vitamin D status during a 12-24 week supervised training program, specifically males and females between the ages of 30 and 50 years old.

DETAILED DESCRIPTION:
Study subjects will be participants in a triathlon training program through the Avera Sports Institute in Sioux Falls, SD. This clinical study will examine changes in iron and vitamin D levels. Blood specimens will be collected at baseline and again after 3 and 6 months of participating in the training program.

ELIGIBILITY:
Inclusion Criteria:

* Males and premenopausal females between the ages of 30 and 50 years old
* Training through the Avera Sports Institute Triathlon Training Program
* Agree to keep diet, exercise and all current health habits stable during participation in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding or planning to become pregnant
* Has a chronic disease that affects calcium or bone metabolism
* Has a chronic disease that affects iron metabolism or iron storage
* Has kidney disease
* Has any laboratory or biometric value that would indicate an issue for the safety of the study subject
* Is currently participating in another clinical research study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and pre-menopausal women between the ages of 30 and 50 who are participating in the Triathlon Training Program through the Avera Sports Institute
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Iron level | baseline, 3 months, 6 months
  Serum iron levels
Vitamin D level | Baseline, 3 months, 6 months
  Serum Vitamin D 25(OH)D levels
C-Reactive Protein level | Baseline, 3 months, 6 months
  Serum C-reactive protein level

SECONDARY OUTCOMES:
Ferritin level | Baseline, 3 months, 6 months
  Serum ferritin level
Hemoglobin level | Baseline, 3 months, 6 months
  Serum hemoglobin level
Hematocrit | Baseline, 3 months, 6 months
  Serum hematocrit level
Total Iron Binding Capacity level | Baseline, 3 months, 6 months
  Serum TBC level

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Vukovich, PhD, Principal Investigator — South Dakota State University
Locations (1):
- Avera Sports Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Gropper SS, Bader-Crowe DM, McAnulty LS, White BD, Keith RE. Non-anemic iron depletion, oral iron supplementation and indices of copper status in college-aged females. J Am Coll Nutr. 2002 Dec;21(6):545-52. doi: 10.1080/07315724.2002.10719253. PMID 12480800
- [Background] Kelley GA, Kelley KS. Effects of aerobic exercise on C-reactive protein, body composition, and maximum oxygen consumption in adults: a meta-analysis of randomized controlled trials. Metabolism. 2006 Nov;55(11):1500-7. doi: 10.1016/j.metabol.2006.06.021. PMID 17046553
- [Background] Malczewska J, Raczynski G, Stupnicki R. Iron status in female endurance athletes and in non-athletes. Int J Sport Nutr Exerc Metab. 2000 Sep;10(3):260-276. doi: 10.1123/ijsnem.10.3.260. PMID 11183845
- [Background] Newhouse IJ, Clement DB. Iron status in athletes. An update. Sports Med. 1988 Jun;5(6):337-52. doi: 10.2165/00007256-198805060-00001. PMID 3041528
- [Background] Okita K, Nishijima H, Murakami T, Nagai T, Morita N, Yonezawa K, Iizuka K, Kawaguchi H, Kitabatake A. Can exercise training with weight loss lower serum C-reactive protein levels? Arterioscler Thromb Vasc Biol. 2004 Oct;24(10):1868-73. doi: 10.1161/01.ATV.0000140199.14930.32. Epub 2004 Jul 29. PMID 15284086
- [Background] Stewart LK, Flynn MG, Campbell WW, Craig BA, Robinson JP, Timmerman KL, McFarlin BK, Coen PM, Talbert E. The influence of exercise training on inflammatory cytokines and C-reactive protein. Med Sci Sports Exerc. 2007 Oct;39(10):1714-9. doi: 10.1249/mss.0b013e31811ece1c. PMID 17909397